CLINICAL TRIAL: NCT04148404
Title: Hypothermic Versus Normothermic Cardiac Bypass in Patients Undergoing CABG Surgery, Effect on Coagulation; Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abdalla, Professor of Anesthesia &I.C.U and Pain Clinic, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Hypothermic vs normothermic
Record Dates: First submitted 2019-10-28; First posted 2019-11-01 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: CABG Surgery, Cold Blood Cardioplegia, Coagulation Profile and Platelet Function

STUDY DESIGN:
Intervention Model Description: Hypothermia may alter coagulation profile of patients undergoing CABG surgery; thus, affecting patients' outcome.
Who Masked: Participant, Care Provider
Masking Description: sealed opaque envelopes prepared by an assistant blinded about the study targets and chosen by patient him/herself, allocated into two groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group NT (Active Comparator): 1.Normothermic group (NT group) included patients will undergo CABG under warm bypass using warm blood cardioplegia (Normothermic CBP).
  Interventions: Procedure: Normothermic group
- Group HT (Active Comparator): 2.Hypothermic group (HT group) included patients will undergo CABG under cold bypass using cold blood cardioplegia (Hypothermic CBP).
  Interventions: Procedure: Normothermic group

INTERVENTIONS:
Procedure: Normothermic group — 1. Normothermic group (NT group) included patients will undergo CABG under warm bypass using warm blood cardioplegia (Normothermic CBP).
  2. Hypothermic group (HT group) included patients will undergo CABG under cold bypass using cold blood cardioplegia (Hypothermic CBP).
  Other Names: Hypothermic group

SUMMARY:
On-pump CABG surgery deleteriously affects hematological and coagulation profiles of patients and this effect was accentuated by the use of cold bypass. PO altered platelet may count and function and prolonged clotting times correlates with amount of daily PO blood wound drainage and number of blood products units used, but prolonged aPTT is the best predictor for these events.

DETAILED DESCRIPTION:
Background: The use of cardiopulmonary bypass during cardiac surgery negatively affects the coagulation system. Hypothermia is also known to inhibit the coagulation profile. The aim of the study is to assess and compare the early postoperative (PO) haematological and coagulation profile of patients undergoing coronary artery bypass graft (CABG) surgery with Hypothermic (HT) versus normothermic (NT) bypass Methods: eighty-six patients were divided into two equal groups: NT group included patients received warm bypass and using warm blood cardioplegia from bypass and HT group included patients received cold bypass and using cold cardioplegia given by the anaesthesiologist. PO monitoring included the activated clotting time (ACT) prior to wound closure and 2-hr changes in the haemoglobin concentration (Hb), platelet count (PC), ADP-induced platelet aggregation (IPA), INR in relation to preoperative profile and amount of PO daily blood loss and number of transfused blood units. The primary outcome was the PO alternations in the coagulation and haematological profile. The secondary outcome was the amount of PO daily bleeding, number of transfused blood units and incidence of re-opening surgery due to bleeding.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic heart disease patients
2. Both genders
3. Aged 50 - 65 years
4. Assigned for first-time, elective and isolated on-pump CABG surgery.

Exclusion Criteria:

1. Pre-existing coagulopathy
2. Hemostasis disorders,
3. Anemia,
4. Redo or emergency CABG, re-exploration for surgical-cause PO bleeding, other associated pathologies, hepatic or renal impairment and/or maintenance on antiplatelet therapy during the last 10 days prior to surgery

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-09 (Actual)

PRIMARY OUTCOMES:
Postoperative alternations in the coagulation and haematological profile | One day Postoperative
  Postoperative alternations in the coagulation and haematological profile

SECONDARY OUTCOMES:
Amount of PO daily bleeding | One day Postoperative
  Amount of PO daily bleeding
Number of transfused blood units | One day Postoperative
  Number of transfused blood units
Incidence of re-opening surgery due to bleeding | 24 hours Postoperative
  Incidence of re-opening surgery due to bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abdalla Mohamed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Till ending our work